CLINICAL TRIAL: NCT03240237
Title: Cardiac Contractility Modulation Therapy in Subjects With Heart Failure With Preserved Ejection Fraction
Brief Title: CCM in Heart Failure With Preserved Ejection Fraction
Acronym: CCM-HFpEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ID_CP_OPT2016-012_0
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure, Diastolic
Keywords: HFpEF
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Intervention Model Description: This pilot study is designed and powered for evaluating the efficacy and safety of CCM therapy in heart failure patients with baseline EF≥50% (HFpEF) who have NYHA Class II or III symptoms despite appropriate medication, for potential expansion of the CE Mark indication for use in the HFpEF population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCM therapy (Experimental): Optimizer SMART
  Interventions: Device: Optimizer SMART

INTERVENTIONS:
Device: Optimizer SMART — Cardiac Contractility Modulation

SUMMARY:
This pilot study will evaluate the efficacy and safety of CCM therapy in heart failure patients with baseline EF≥50% (HFpEF) who have New York Heart Association (NYHA) Class II or III symptoms despite appropriate medication.

The terminology of the HF classification HFpEF is based on the 2016 European Society of Cardiology (ESC) Heart Failure Guidelines.

DETAILED DESCRIPTION:
This is a pilot clinical study of CCM in addition to optimal medical therapy (OMT) over a 24 week period.The primary endpoint shall be mean change from baseline to 24 weeks in Kansas City Cardiomyopathy Questionnaire (KCCQ) overall score (reflecting integrated information on physical limitations, symptoms, self-efficacy, social interference and quality of life).

This pilot study will collect efficacy and safety data in heart failure patients having NYHA class II and III symptoms despite appropriate medication with baseline ejection fraction equal or greater than 50% (HFpEF populations).

ELIGIBILITY:
1. Inclusion criteria

   1. Baseline ejection fraction ≥ 50% (as assessed by echocardiogram within 30 days of enrollment and confirmed by the echo core laboratory).
   2. NYHA class II or III symptoms despite receiving stable optimal medical therapy (OMT) for at least 30 days based on patient's medical records (chronic stable, not transient or crescendo heart failure or angina pectoris)
   3. Stable optimal medical therapy for Heart failure for 3 months.
   4. NT-proBNP > 220 pg/ml for subjects in sinus rhythm or > 600 pg/ml for subjects in atrial fibrillation
   5. Has the following (as assessed by the core lab):

      * LAVi ≥ 34 ml/m² or LVH >12mm AND either
      * E/e' ≥ 13 OR
      * septal e' < 7 cm/s or lateral e' <10 cm/s
   6. Patient giving informed consent, willing to be available for scheduled study follow-up visits, and able to complete all testing of the study protocol
2. Exclusion criteria

   1. Age below 40 or greater than 80
   2. Patients with expected lifespan of less than 12 months from time of enrollment
   3. Subjects referred to an institution based on a judicial or administrative order
   4. Dilated left ventricle, as evidenced by LVEDVI >= 97 mL/m2 (as assessed by the echo core lab)
   5. Primary cardiac valvular disease (anything more than grade 2)
   6. Congenital or untreated ischemic heart disease
   7. Infiltrative / inflammatory / genetic cardiomyopathy as documented in the medical record (e.g. amyloid, hemochromatosis, myocarditis, hypertrophic cardiomyopathy, M. Fabry, cardiac tumor), or persistent large pericardial effusion
   8. Unstable or frequent (>1 episode/week) angina pectoris
   9. Hospitalization for HF requiring the use of inotropic support or IABP within 30 days of enrollment
   10. Systolic Blood Pressure > 160 mmHg
   11. Uncorrected severe anemia (e.g. hemoglobin <9g/dL)
   12. PR interval greater than 375 ms
   13. Exercise tolerance limited due to noncardiac disorders (e.g. deconditioning, severe lung disease, frailty)
   14. Scheduled for a cardiac surgery or a PCI procedure, or had a cardiac surgery procedure within 90 days or a PCI procedure within 30 days prior to enrollment
   15. Myocardial infarction within 90 days of enrollment
   16. Cardioversion within 30 days of enrollment
   17. History of significant ectopy either on 12-lead ECG or Holter monitoring (more than 10% PVCs).
   18. Heart rate > 110 bpm on ECG for patients with atrial fibrillation
   19. Mechanical tricuspid valve
   20. Prior heart transplant or ventricular assist device
   21. Pregnant or planning to become pregnant during the study
   22. Breastfeeding subjects
   23. Subject participating in another medical therapy or device related study, unrelated to CCM™, at the same time or within 30 days prior to enrollment into this study
   24. Subjects on dialysis, or with documented GFR<30 or with other major medical disorder (e.g. severe anemia, liver failure)
   25. Subjects with any active non-cardiac implants

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
KCCQ change | 24 weeks
  Mean change from baseline to 24 weeks in Kansas City Cardiomyopathy Questionnaire (KCCQ) overall score

SECONDARY OUTCOMES:
Echocardiography | 24 weeks
  LAVi and diastolic function: septal E' velocity, septal E/E' ratio
NT-proBNP | 24 weeks
  Mean Change in 24 weeks
NYHA class | 24 weeks
  Mean Change in 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Tschoepe, Prof., Principal Investigator — University Hospital Charite Berlin
Locations (17):
- Australia (3):
  - Friendly Society Private Hospital, Bundaberg, Queensland
  - St. John of God Bunbury, Bunbury
  - St. John of God Murdoch Hospital, Perth
- Hospital Na Homolce, Prague, Czechia
- Kerckhoff-Klinik GmbH, Bad Nauheim, Hesse, Germany
- Italy (3):
  - INRCA IRCCS Ancona, Ancona, Rome
  - Auxologico Institute, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego zakład leczniczy Centralnego Szpitala Klinicznego, Warsaw
  - Uniwersytecki Szpital Kliniczny we Wrocław, Wroclaw
  - 4 Wojskowy Szpital Kliniczny z Poliklinika SPZOZ we Wroclawiu, Wroclaw
- West Lisbon Hospital Center, E.P.E., hereinafter referred to as CHLO, E.P.E, Lisbon, Portugal
- Spain (4):
  - Santiago de Compostella -- Servicio de Cardiología y UCC/ Cardiology and Coronary Care Department Hospital Clínico Universitario. XXI de Santiago de Compostela SERGAS, Santiago de Compostela, C/ A Choupana S.n
  - Hospital General de Alicante, Alicante
  - Hospital Universitario 12 de Octubre Unidad de Insuficiencia Cardiaca y Trasplante Servicio de Cardiología, Planta 6. Bloque D.Ciber 8, Madrid
  - Hospital Alvaro Cunquero, Vigo
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tschope C, Van Linthout S, Spillmann F, Klein O, Biewener S, Remppis A, Gutterman D, Linke WA, Pieske B, Hamdani N, Roser M. Cardiac contractility modulation signals improve exercise intolerance and maladaptive regulation of cardiac key proteins for systolic and diastolic function in HFpEF. Int J Cardiol. 2016 Jan 15;203:1061-6. doi: 10.1016/j.ijcard.2015.10.208. Epub 2015 Oct 27. No abstract available. PMID 26638055
- [Result] Linde C, Grabowski M, Ponikowski P, Rao I, Stagg A, Tschope C. Cardiac contractility modulation therapy improves health status in patients with heart failure with preserved ejection fraction: a pilot study (CCM-HFpEF). Eur J Heart Fail. 2022 Dec;24(12):2275-2284. doi: 10.1002/ejhf.2619. Epub 2022 Aug 11. PMID 35855646